CLINICAL TRIAL: NCT05235061
Title: HOme-Based Self-management and COgnitive Training CHanges Lives (HOBSCOTCH) -Post-Traumatic Epilepsy (PTE)
Acronym: HOBSCOTCHPTE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Barbara Jobst, Chair, Department of Neurology; Professor of Neurology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY02001238; W81XW82110279 (Other: US Department of Defense)
Record Dates: First submitted 2022-01-11; First posted 2022-02-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy, Traumatic; Brain Injuries, Traumatic
Keywords: Epilepsy; Epilepsy, Post-Traumatic; Traumatic Brain Injury; Cognition; Self-Management; Cognitive remediation; Seizures; Memory Disorders; Caregivers; Caregiver Burden; Mindfulness
MeSH Terms: conditions — Epilepsy, Post-Traumatic; Brain Injuries, Traumatic; Epilepsy; Seizures; Memory Disorders; Caregiver Burden | interventions — Caregivers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PTE Participant Group 1 (Experimental): PTE Participant Group 1 will receive the HOBSCOTCH-PTE intervention consisting of 1:1 sessions delivered once per week including:
  * 1 pre-HOBSCOTCH Session (on webcam)
  * 1 educational session (on webcam)
  * 6 telephone sessions
  * 1 wrap-up session (webcam or telephone)
  Interventions: Behavioral: Home Based Self-management and Cognitive Training Changes lives in post traumatic epilepsy (HOBSCOTCH-PTE)
- PTE Participant Group 2 (Other): PTE Participant Group 2 will be on a 3-month wait list after which they will receive HOBSCOTCH-PTE consisting of 1:1 sessions delivered once per week including:
  * 1 pre-HOBSCOTCH Session (on webcam)
  * 1 educational session (on webcam)
  * 6 telephone sessions
  * 1 wrap-up session (webcam or telephone)
  Interventions: Behavioral: Home Based Self-management and Cognitive Training Changes lives in post traumatic epilepsy (HOBSCOTCH-PTE)
- PTE Caregiver Group 1 (Experimental): Caregiver Group 1 will receive an adapted version of HOBSCOTCH-PTE by attending session 1 of the HOBSCOTCH-PTE (virtual) program with their PTE patient as well as guidance and instructions on utilizing quick relaxation. Caregiver Group 1 will also attend session 8 of the program with the PTE patient to focus on program wrap-up and maintenance planning.
  Interventions: Behavioral: HOBSCOTCH-PTE for Caregivers
- PTE Caregiver Group 2 (Other): Caregiver Group 2 will be on a 3 month wait list with their PTE patient after which time they will receive an adapted version of HOBSCOTCH-PTE by attending session 1 of the HOBSCOTCH-PTE (virtual) program with their PTE patient as well as guidance and instructions on utilizing quick relaxation. Caregiver Group 2 will also attend session 8 of the program with the PTE patient to focus on program wrap-up and maintenance planning.
  Interventions: Behavioral: HOBSCOTCH-PTE for Caregivers

INTERVENTIONS:
Behavioral: Home Based Self-management and Cognitive Training Changes lives in post traumatic epilepsy (HOBSCOTCH-PTE) — HOBSCOTCH is a home-based self-management program to treat cognitive symptoms and improve quality of life, while minimizing the barriers of access to care. The program is based on Problem Solving Therapy (PST) and teaches problem solving strategies and compensatory mechanisms to help manage cognitive dysfunction and enhance quality of life. HOBSCOTCH-PTE is an adaptation of the HOBSCOTCH program for people with a traumatic brain injury and post-traumatic epilepsy that incorporates education about TBI, PTE, and cognition into the education module.
  Other Names: HOBSCOTCH-PTE
  Arms: PTE Participant Group 1; PTE Participant Group 2
Behavioral: HOBSCOTCH-PTE for Caregivers — Select components of the HOBSCOTCH-PTE program delivered to caregivers consist of session 1 of the HOBSCOTCH-PTE (virtual) program (education module), guidance and instructions on utilizing quick relaxation, and session 8 of the HOBSCOTCH-PTE program (program wrap-up and maintenance planning).
  Arms: PTE Caregiver Group 1; PTE Caregiver Group 2

SUMMARY:
The purpose of this study is to assess the ability of the home-based intervention, HOBSCOTCH-PTE, to improve the quality of life and cognitive function in Service Members, Veterans and civilians with post traumatic epilepsy (PTE). This study will also assess the ability of the HOBSCOTCH-PTE program to improve quality of life in caregivers of PTE patients and to reduce caregiver burden.

DETAILED DESCRIPTION:
The investigators hypothesis is that the home-based intervention (HOBSCOTCH-PTE) will improve quality of life and cognitive function in Service Members, Veterans and civilians with PTE. The integration of family caregiver participation in the HOBSCOTCH-PTE intervention will reduce caregiver burden and increase caregiver knowledge of their loved one's disease and cognitive challenges they face, ultimately leading to an improvement in caregiver quality of life.

The investigators will test the hypothesis by pursuing the following specific aims:

Aim 1: Adapt the HOBSCOTCH program education module for delivery to patients with PTE and cognitive challenges. The investigators working hypothesis is that the existing education module of the HOBSCOTCH program can be adapted to address key knowledge areas for patients with TBI and PTE and their caregivers.

Aim 2: Evaluate the efficacy of the HOBSCOTCH-PTE program in patients with PTE. The investigators working hypothesis is that the HOBSCOTCH-PTE intervention will improve QOL in PTE patients. The investigators also expect to see improvements in subjective cognition, knowledge, self-efficacy, symptom reduction, and health outcomes.

Aim 3: Incorporate family caregivers into select components of the HOBSCOTCH-PTE intervention and evaluate the effects of the HOBSCOTCH-PTE intervention on the caregiver. The investigators working hypothesis is that family caregivers will have improvement in QOL, caregiver burden, and health status as a result of their family member with PTE participating in the HOBSCOTCH-PTE intervention, and by their own participation in the HOBSCOTCH-PTE modules delivering disease specific education and mindfulness skill building exercises.

ELIGIBILITY:
Inclusion Criteria/PTE Participants:

* Age 18+
* Diagnosis of post traumatic epilepsy, with controlled or uncontrolled seizures
* Subjective memory complaints
* No changes in antiepileptic and antidepressant medication regimen for 1 month, however brief discontinuation of antiepileptic medicine for inpatient video EEG evaluation is acceptable
* Literate and proficient in English
* Telephone access
* Internet access

Exclusion Criteria/PTE Participants:

* Subjects self-reporting a dementing illness or a mention of a dementing illness in their medical record
* Severe mental disability or estimated IQ less than 70 per clinical judgement
* Significant visual impairment precluding reading or writing
* No reliable telephone or internet access
* No diagnosis of epilepsy

Inclusion Criteria/Caregiver Participants

* Age 18+
* Caregivers to a patient with a confirmed diagnosis of PTE
* Literate and proficient in English
* Telephone access
* Internet access

Exclusion Criteria/Caregiver Participants:

* Significant visual impairment precluding reading or writing
* No reliable telephone or internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life as measured by comparing QOLIE-31 scores at baseline and 3 months post-intervention in participants with PTE | Baseline and 3 months post-intervention.
  The Quality of Life in Epilepsy (QOLIE-31) is a validated tool containing 16 multi-item scales which assess health related quality of life, emotional well-being, memory and attention deficits, medication effects, seizure control, psychosocial functioning, and health perception. Scores range from 0 to 100, with a higher score reflecting a higher quality of life.
Change in subjective cognition as measured by comparing NeuroQOL - Cognitive Function sub-scale scores at baseline and 3 months post-intervention in participants with PTE | Baseline, 3 months, 6 months
  The Cognitive Function sub-scale of the NeuroQOL is a brief validated tool developed by the NIH for use in patients with neurological disease. Scores range from 8 to 40, with a higher score indicating better reported cognitive functioning.
Change in caregiver burden as measured by comparing Zarit Burden Interview scores at baseline and at 3 months post-intervention in caregivers of PTE participants | Baseline and 3 months post-intervention
  The Zarit Burden Interview is a 22-item questionnaire designed to measure the extent to which a caregiver perceives his or her level of burden as a result of caring for a person with a particular diagnosis. A 5 point Likert scale is used with a higher score indicating a greater level of perceived burden.

SECONDARY OUTCOMES:
Changes in PTE participant knowledge of their own epilepsy as measured by comparing scores on the Epilepsy Knowledge of Own Condition questionnaire at baseline and 6 months post-intervention. | Baseline and 6 months post-intervention.
  The Epilepsy Knowledge of Own Condition is a 23 item, mostly YES/NO, questionnaire developed and validated by S. Jarvie, C. Espie, M. Brodie Published 1 September 1993questionnaire to assess knowledge of epilepsy: 2-knowledge of own condition.
Changes in PTE participants self-efficacy (subjective impression of managing their life with epilepsy) as measured by comparing scores on the Epilepsy Self-Efficacy Scale at baseline and at 3 months post-intervention. | Baseline and 3 months post-intervention.
  The Epilepsy Self-Efficacy Scale is validated a 33-item scale that measures the different aspects of efficacy in the self-management of epilepsy. Items are rated on an 11-point Likert rating scale, ranging from 0, I cannot do at all, to 10, sure I can do.
Changes in PTE participants' objective cognition as measured by comparing scores on the Montreal Cognitive Assessment (MoCA) at baseline and at 3 months post-intervention. | Baseline and 3 months post-intervention.
  The Montreal Cognitive Assessment (MoCA) is a validated 30 item test that helps healthcare professionals detect cognitive impairments.
Changes in PTE Participants' mood as measured by comparing scores on the Patient Health Questionnaire (PHQ-9) at baseline and at 3 months post- intervention. | Baseline and at 3 months post-intervention
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Changes in seizure frequency (PTE participants) as measured by comparing daily self-reported seizures at baseline and at 3 months post-intervention | Recorded daily and compared between baseline and 3 months-post intervention.
  PTE participants will self-report their seizure activity using a smartphone app or paper log. The smart phone app was developed by the HOBSCOTH program at Dartmouth-Hitchcock and is used clinically in the HOBSCOTCH program.
Changes in PTE participants' medication adherence as measured by a daily self-reported diary compared at baseline and at 3 months post-intervention. | Recorded daily and compared between baseline and 3 months post-intervention.
  PTE participants will self-report their medication adherence activity using a smartphone app or paper log. The smart phone app was developed by the HOBSCOTH program at Dartmouth-Hitchcock and is used clinically in the HOBSCOTCH program.
Changes in PTE participants' use of memory strategies as measured by a daily self-reported diary compared at baseline and 3 months post-intervention. | Recorded daily and compared between baseline and 3 months post-intervention.
  PTE participants will self-report their use of the memory strategies they learn in the HOBSCOTCH-PTE program using a smartphone app developed by the HOBSCOTH program at Dartmouth-Hitchcock or in a paper log.
Changes in PTE participants' self-reports of wellbeing as measured by comparing daily reports of well-being in a diary at baseline and at 3 months post-intervention. | Recorded daily and compared between baseline and 3 months post-intervention.
  The researchers will collect daily well-being information throughout the entire study by use of a smartphone app or paper log and a basic single item Likert-scale of well-being.
Changes in Caregiver Participants' knowledge of epilepsy as measured by comparing scores on the [Caregiver] General Knowledge of Epilepsy questionnaire at baseline and at 6 months-post intervention. | Baseline and 6 months post-intervention.
  The [Caregivers] General Knowledge of Epilepsy is a validated 34 item TRUE/FALSE questionnaire developed to assess general knowledge of epilepsy. (Jarvie S, Espie CA, Brodie MJ. The development of a questionnaire to assess the knowledge of epilepsy, 1: general knowledge of epilepsy. Seizure 1993; 2: 179- 85.)
Changes in caregiver self-reported health status as measured by comparing scores on the Short-Form 36 (SF-36) at baseline and 3 months-post intervention. | Baseline and 3 months post-intervention.
  The Short Form Health Survey (SF-36) is a validated 36-item, patient-reported survey of patient health. It consists of 8 sub-scales, which are scored on a 3-point, 5-point or dichotomous (yes/no or true/false) scale. The scores are converted to a 1 - 100 point scale with a lower score indicating more disability, i.e. 0 = maximum disability and 100 = no disability.
Changes in Caregiver Participants' mood as measured by comparing scores on the Patient Health Questionnaire (PHQ-9) at baseline and at 3 months post- intervention. | Baseline and at 3 months post-intervention
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Sustainability of improvement on primary outcome measure for PTE Participants by comparing scores on the QOLIE-31 at 3 months and 6 months post-intervention. | 3 months 6 months post intervention.
  The Quality of Life in Epilepsy (QOLIE-31) is a validated tool containing 16 multi-item scales which assess health related quality of life, emotional well-being, memory and attention deficits, medication effects, seizure control, psychosocial functioning, and health perception. Scores range from 0 to 100, with a higher score reflecting a higher quality of life.
Sustainability of improvement on primary outcome measures for PTE Participants by comparing scores on the Cognitive Function sub-scale of the NeuroQOL at 3 months and 6 months post-intervention. | 3 months 6 months post intervention.
  The Cognitive Function sub-scale of the NeuroQOL is a brief validated tool developed by the NIH for use in patients with neurological disease. Scores range from 8 to 40, with a higher score indicating better reported cognitive functioning.
Sustainability of improvement on primary outcome measures for Caregiver Participants by comparing scores on the Zarit Caregiver Burden at 3 months and 6 months post-intervention. | 3 months 6 months post intervention.
  The Zarit Burden Interview is a 22-item questionnaire designed to measure the extent to which a caregiver perceives his or her level of burden as a result of caring for a person with a particular diagnosis. A 5 point Likert scale is used with a higher score indicating a greater level of perceived burden.
Engagement and Satisfaction for PTE Participants as measured by analyzing study attrition and a Participant Satisfaction Survey at the end of the study. | 6 months post-intervention (end of study)
  The Participant Satisfaction Survey has been developed through the original HOBSCOTH program and is used in clinical practice for quality improvement. It contains 10 items scored on a 5-point Likert scale with a higher score indicating greater satisfaction with the program.
HOBSCOTCH Fidelity and Compliance as measured by completed sessions and completed homework for PTE Participants. | 6 months post-intervention (end of study)
  Completed sessions and homework are tracked throughout the study by the certified HOBSCOTCH coaches.
Feasibility of HOBSCOTCH program for Caregivers as measured by study attrition and a Participant Satisfaction Survey. | 6 months post-intervention (end of study)
  The Participant Satisfaction Survey was developed through the original HOBSCOTH program and is used in clinical practice for quality improvement. It has been modified to address Caregiver's satisfaction as a result or participating in this study and contains 9 items scored on a 5-point Likert scale with a higher score indicating greater satisfaction with the program.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara C. Jobst, MD, Dr. Med., Principal Investigator — Dartmouth-Hitchcock Medical Center; Elaine T Kiriakopoulos, MD, MSc, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dartmouth-Hitchcock study team will share data with the MEW Network Database team at Case Western Reserve University. HOBSCOTCH is a part of the Managing Epilepsy Well Network (MEWN), MEWN has been a national leader in developing, testing and disseminating evidence-based epilepsy self-management programs. Collectively, the MEWN has an integrated database using MEW common data elements (e.g., demographics, seizure details, quality of life, depression) (1).
  Sajatovic, M., B. Wilson, R. Shegog, B.S.B. F, C. Escoffery, B.C. Jobst, E.K. Johnson, R.T. Fraser, R.C. Quarells, and T.M. Spruill, The Managing Epilepsy Well (MEW) network database: Lessons learned in refining and implementing an integrated data tool in service of a national U.S. Research Collaborative. Epilepsy Behav, 2021. 115: p. 107650.
Supporting Information: Study Protocol
Time Frame: conclusion of study
Access Criteria: The Dartmouth-Hitchcock study team will work directly with the MEW Network Database team at Case Western Reserve University; a current data sharing plan is in place.

REFERENCES:
- [Background] Caller TA, Ferguson RJ, Roth RM, Secore KL, Alexandre FP, Zhao W, Tosteson TD, Henegan PL, Birney K, Jobst BC. A cognitive behavioral intervention (HOBSCOTCH) improves quality of life and attention in epilepsy. Epilepsy Behav. 2016 Apr;57(Pt A):111-117. doi: 10.1016/j.yebeh.2016.01.024. Epub 2016 Mar 2. PMID 26943948